CLINICAL TRIAL: NCT00718614
Title: Choroidal Blood Flow Changes During Dark/Light Transitions in Patients With IDDM
Brief Title: Choroidal Blood Flow Changes During Dark/Light Transitions in Patients With Insulin-dependent Diabetes Mellitus (IDDM)
Status: Terminated | Phase: Not Applicable | Type: Interventional
Sponsor: Medical University of Vienna (Other)
Responsible Party: Principal Investigator, Gerhard Garhofer, Assoc. Prof. Priv. - Doz. Dr, Medical University of Vienna
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Basic Science
Other Study IDs: OPHT-300505-2
Record Dates: First submitted 2008-07-07; First posted 2008-07-18 (Estimated); Last update posted 2014-11-25 (Estimated); Status verified 2014-11

CONDITIONS: Diabetes Mellitus, Type 1; Diabetic Retinopathy
Keywords: Choroidal blood flow; Laser Doppler flowmetry; Diabetic Retinopathy; Diabetic Neuropathy
MeSH Terms: conditions — Diabetes Mellitus, Type 1; Diabetic Retinopathy; Diabetic Neuropathies

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (4):
- 1 (Other): Patients with long standing IDDM (>10 years) and no diabetic retinopathy
  Interventions: Procedure: Light will be switched from 0.5µW/cm2/sr to 115µW/cm2/sr.
- 2 (Other): Patients with long standing IDDM (>10 years) and mild non-proliferative diabetic retinopathy
  Interventions: Procedure: Light will be switched from 0.5µW/cm2/sr to 115µW/cm2/sr.
- 3 (Other): Patients with long standing IDDM (>10 years) and moderate to severe non-proliferative diabetic retinopathy
  Interventions: Procedure: Light will be switched from 0.5µW/cm2/sr to 115µW/cm2/sr.
- 4 (Other): healthy volunteers, matched for age and sex
  Interventions: Procedure: Light will be switched from 0.5µW/cm2/sr to 115µW/cm2/sr.

INTERVENTIONS:
Procedure: Light will be switched from 0.5µW/cm2/sr to 115µW/cm2/sr. — Light will be switched from 0.5µW/cm2/sr to 115µW/cm2/sr.

SUMMARY:
There is evidence from a variety of animal studies that choroidal blood flow is under neural control. Recent results in humans indicate that a light/dark transition is associated with a short lasting reduction in choroidal blood flow. Several observations indicate that the changes in choroidal perfusion are triggered at least in part by neural mechanisms. Particularly, we have shown that during unilateral dark/light transition both eyes react with choroidal vasoconstriction strongly indicating a neural mechanism for blood flow regulation. Investigation of changes in choroidal blood flow during light/dark transition may represent an interesting approach to study neural dysregulation at the level of the eye in patients with IDDM. Accordingly, the hypothesis of reduced choroidal blood flow responses to a light/dark transition in patient with IDDM will be tested. This response in choroidal blood flow will be correlated to parameters of diabetic neuropathy and diabetic retinopathy.

ELIGIBILITY:
Inclusion Criteria:

For healthy control subjects:

* Men and women aged over 18 years, matched in regard to age, sex and smoking status
* Normal findings in the medical history and physical examination unless the investigator considers an abnormality to be clinically irrelevant
* Normal laboratory values unless the investigator considers an abnormality to be clinically irrelevant
* Normal ophthalmic findings, Ametropia < 3 dpt for healthy control subjects

For patients with IDDM:

* Men and women aged over 18 years
* Normal findings in the medical history and physical examination unless the investigator considers an abnormality to be clinically irrelevant
* Long standing IDDM > 10 years
* Mild or moderate to severe non-proliferative diabetic retinopathy (defined according to the MAHC)
* Ametropia < 3 dpt

Exclusion Criteria:

Any of the following will exclude a healthy subject from the study:

* Regular use of vasoactive medication with may interfere with the study procedure, abuse of alcoholic beverages, participation in a clinical trial in the 3 weeks preceding the study
* Symptoms of a clinically relevant illness in the 3 weeks before the first study day
* Blood donation during the previous 3 weeks

Any of the following will exclude a patient with IDDM from the study:

* Evidence of any relevant retinal or choroidal disease (Glaucoma, age related macula degeneration, cataract, history of central retinal artery obstruction or central retinal vein thrombosis)
* Ophthalmological surgery (history of photo laser coagulation, including argon laser trabeculoplasty (ALT), trabeculectomy, deep sclerectomy)
* History of intravitreal injection with anti-proliferative therapy
* Need for dialysis
* Non-treated systemic hypertension (SPB>150, DBP>95)
* Evidence of coronary heart disease, cardiomyopathy, stenocardia, congestive heart failure, peripheral occlusive vascular disease, cardiac autonomic neuropathy
* Symptoms of a clinically relevant illness in the 3 weeks before the first study day
* Blood donation during the previous 3 weeks

Min Age: 19 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 80 (Estimated)
Dates: Start 2007-06; Primary Completion 2007-07 (Actual); Study Completion 2007-07 (Actual)

PRIMARY OUTCOMES:
fundus pulsation amplitude | 3 hours
choroidal blood flow | 3 hours

SECONDARY OUTCOMES:
Nerve conduction velocity | measured before intervention
Pupil diameter during infra-red pupillometry | measured before intervention
heart rate variability | measured before intervention

CONTACTS AND LOCATIONS:
Overall Officials: Gerhard Garhoefer, MD, Principal Investigator — Department of Clinical Pharmacology, Medical University of Vienna
Locations (1):
- Department of Clinical Pharmacology, Vienna, Austria